CLINICAL TRIAL: NCT01295853
Title: T3 Versus T4 Sympathicotomy for Treatment of Primary Palmar Hyperhidrosis: a Prospective Randomized Study
Brief Title: T3 Versus T4 Sympathicotomy for Treatment of Primary Palmar Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: dr. ahmed negm, manoura university hospial
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMRO2345
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Compensatory Hyperhidrosis; Recurrence
MeSH Terms: conditions — Recurrence | interventions — Sympathectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- t3 sympathicotomy (Active Comparator): The sympathetic chain was identified at the level of the crossing of the third or fourth costal heads after dissection of the parietal pleura and completely divided about 1 cm wide at the upper margin of the rib. With assistance of anaesthesia team we reinflate the lung totally in sequence with removal of the trocars. The same procedure was performed on the opposite side and ablation of the sympathetic chain overlying the rib was performed bilaterally. At the end of surgery, a postoperative chest x-ray was routinely taken to rule out pneumothorax or hemothorax.
  Interventions: Procedure: t3 sympathicotomy; Procedure: t4 symapthicotomy
- t4 sypathicotomy (Active Comparator): The sympathetic chain was identified at the level of the crossing of the third or fourth costal heads after dissection of the parietal pleura and completely divided about 1 cm wide at the upper margin of the rib. With assistance of anaesthesia team we reinflate the lung totally in sequence with removal of the trocars. The same procedure was performed on the opposite side and ablation of the sympathetic chain overlying the rib was performed bilaterally. At the end of surgery, a postoperative chest x-ray was routinely taken to rule out pneumothorax or hemothorax.
  Interventions: Procedure: t4 symapthicotomy

INTERVENTIONS:
Procedure: t3 sympathicotomy — The sympathetic chain was identified at the level of the crossing of the third or fourth costal heads after dissection of the parietal pleura and completely divided about 1 cm wide at the upper margin of the rib. With assistance of anaesthesia team we reinflate the lung totally in sequence with removal of the trocars. The same procedure was performed on the opposite side and ablation of the sympathetic chain overlying the rib was performed bilaterally. At the end of surgery, a postoperative chest x-ray was routinely taken to rule out pneumothorax or hemothorax.
  Other Names: sympathectomy
  Arms: t3 sympathicotomy
Procedure: t4 symapthicotomy — The sympathetic chain was identified at the level of the crossing of the third or fourth costal heads after dissection of the parietal pleura and completely divided about 1 cm wide at the upper margin of the rib. With assistance of anaesthesia team we reinflate the lung totally in sequence with removal of the trocars. The same procedure was performed on the opposite side and ablation of the sympathetic chain overlying the rib was performed bilaterally. At the end of surgery, a postoperative chest x-ray was routinely taken to rule out pneumothorax or hemothorax.
  Other Names: sympathectomy

SUMMARY:
T3 versus T4 as a primary treatment for palmer hyperhydrosis and effect on postoperative compensatory hyperhydrosis

DETAILED DESCRIPTION:
Palmar hyperhidrosis (PH) is a benign sympathetic disorder that does not threaten health but affects daily activities, and may causes social withdrawal and even depression.1 An incidence of up to 1% has been reported by various series in the literature. The incidence in men and women is the same; however women are more likely to seek medical attention, which may explain the higher incidence of female patients in most surgical series [2,3]. Although various treatment options are available, including topical and systemic therapies, iontophoresis, regional nerve block, and botulinum toxin injection, each has its limitations 4. Video-assisted thoracoscopic sympathetic surgery is currently a worldwide accepted treatment of primary palmar hyperhidrosis (PH) 5. However, compensatory hyperhidrosis (CH) is the most common and serious side effect that occurs in 30-70% of patients after T2 or T2-3 sympathectomy 6. For that now T2 sympathetic surgeries are seldom used in PH. Procedures that involve T3 or/and T4 sympathetic ganglions are widely accepted in many centers with favourable results.5 But some patients still present with certain degrees of CH or over dry hands after operation 7, 8.

The aim of this study is to compare the two methods for the treatment of PH, in which the sympathetic chain was transected in merely one segment, on the level of either the third or the fourth ribbed, defined as T3 sympathicotomy or T4 sympathicotomy, respectively. Emphasis was placed on the evaluation of the efficacy, side effects, and patients' satisfaction rate to these two types of surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary palmar hyperhidrosis

Exclusion Criteria:

* Patients with pleural adhesion
* Bleeding diathesis
* Local infection
* Patients with certain anatomic anomalies

Ages: 15 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
postoperative compensatory hyperhidrosis | 2008-2010
  CH remains the most common and distressing complication postsympathicotomy and many efforts have been made to ovoid its happening .Chou et al, 2 suggested that the underlying mechanism of CH may be due to a reflex response in sweating centre in hypothalamus but the exact mechanism beyond this phenomenon remain unclear.

SECONDARY OUTCOMES:
improvement of planter sweating assessment of overdry hands early postoperative complication ( pneumothorax,,,,,) recurrance | 2008-2010
  The recurrence rate in T4 group was occurring in 2 patients (2.8%), whereas one recurrence found in T3 group (1.5%).
  Kim et al 4, reported a 4.2 % of patients undergo T3 sympathicotomy complaining of gustatory sweating in a study carried out on 56 patients. However In our study there was no occurrence of postsympathicotomy gustatory hyperhidrosis and this may be due to the small numbers in our series.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed negm, md, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Background] Chou SH, Kao EL, Lin CC, Chang YT, Huang MF. The importance of classification in sympathetic surgery and a proposed mechanism for compensatory hyperhidrosis: experience with 464 cases. Surg Endosc. 2006 Nov;20(11):1749-53. doi: 10.1007/s00464-005-0829-7. Epub 2006 Oct 5. PMID 17024534